CLINICAL TRIAL: NCT02403856
Title: Efficacy and Tolerance of Ultrasound-guided Needling and Lavage of Calcific Tendinitis of the Rotator Cuff Performed With or Without Subacromial Corticosteroid Injection: A Double Blind Controlled Study
Brief Title: Efficacy and Tolerance of Ultrasound-guided Needling and Lavage of Calcific Tendinitis of the Rotator Cuff Performed With or Without Subacromial Corticosteroid Injection
Acronym: CALCECHO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC15_0019
Record Dates: First submitted 2015-03-20; First posted 2015-03-31 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Calcifying Tendinitis of Shoulder
Keywords: calcifying tendinitis; Needle lavage; Shoulder; Corticosteroid injection; Ultrasound-guided
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy | interventions — Sodium Chloride; Methylprednisolone Acetate; Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Sodium Chloride 0.9%) (Experimental): Needling and lavage of calcific tendinitis of the rotator cuff followed by the injection of sterile physiological Saline (Sodium Chloride 0.9%) in the subacromial bursae.
  Interventions: Drug: Sodium Chloride 0.9%; Procedure: Ultrasound-guided Needling and Lavage
- Control group (Methylprednisolone Acetate) (Active Comparator): Needling and lavage of calcific tendinitis of the rotator cuff followed by the injection of methylprednisolone acetate in the subacromial bursae
  Interventions: Drug: Methylprednisolone acetate; Procedure: Ultrasound-guided Needling and Lavage

INTERVENTIONS:
Drug: Sodium Chloride 0.9% — Needling and lavage of calcific tendinitis of the rotator cuff followed by the injection of sterile physiological Saline (Sodium Chloride 0.9%) in the subacromial bursae.
  Other Names: NaCl 0.9%
  Arms: Experimental group (Sodium Chloride 0.9%)
Drug: Methylprednisolone acetate — Needling and lavage of calcific tendinitis of the rotator cuff followed by the injection of methylprednisolone acetate in the subacromial bursae
  Other Names: Dépomédrol
  Arms: Control group (Methylprednisolone Acetate)
Procedure: Ultrasound-guided Needling and Lavage

SUMMARY:
Calcific tendinitis of the rotator cuff is a common cause of chronic pain of the shoulder. Needling and lavage of the calcification is one of the therapeutic options after failure of conservative management with physiotherapy and anti-inflammatory drugs. Needling is usually followed by a corticosteroid injection in the subacromial bursae in order to prevent acute pain reaction due to the intervention. However, the relevance of this injection has never been proven. Moreover, corticosteroid could prevent the inflammatory reaction induced by the needling and thus the body's natural calcium resorption processes. Finally, corticosteroids could have deleterious effect on the tendon structures and favour local infection. Our hypothesis is that corticosteroid have no significant effect on acute pain after needling and therefore should not been performed systematically after needling.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain for at least 3 month
* Positive Hawkins, Yocum and/or Neer test for impingement
* Calcific deposit >= 5 mm on shoulder x-ray in one the tendon of the rotator cuff

Exclusion Criteria:

* Allergy to lidocaïne or methylprednisolone acetate
* Acute pain suggestive of resorption of the calcification with ill-defined - calcification on X-Ray
* Other shoulder diseases : ostearthritis of the gleno-humeral or acromio-clavicular joint
* Sonographic findings of rotator cuff tear
* Subacromial steroid injection in the previous month
* Uncontrolled diabetes
* Pregnant women
* Contraindication for the use of nonsteroidal antiinflammatory drugs or paracetamol/acetaminophene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-04-04 (Actual); Primary Completion 2017-04-02 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Maximum pain (VAS scale) | 7 days
  Maximum pain on a VAS scale (0-10) reported by the patient in the seven days following the needling.

SECONDARY OUTCOMES:
Anti-inflammatory and analgesic intake | 7 days
Size of the calcific deposit | 7 days
Size of the calcific deposit | 3 months
Size of the calcific deposit | 12 months
Number of frozen shoulder in each group | 7 days
Number of frozen shoulder in each group | 6 weeks
Number of frozen shoulder in each group | 3 months
Number of frozen shoulder in each group | 6 months
Number of frozen shoulder in each group | 12 months
VAS pain during daily activity | 7 days
VAS pain during daily activity | 6 weeks
VAS pain during daily activity | 3 months
VAS pain during daily activity | 6 months
VAS pain during daily activity | 12 months
VAS pain at rest | 7 days
VAS pain at rest | 6 weeks
VAS pain at rest | 3 months
VAS pain at rest | 6 months
VAS pain at rest | 12 months
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | 7 days
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | 6 weeks
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | 3 months
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | 6 months
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - La Roche sur Yon Hospital, La Roche-sur-Yon
  - Nantes University Hospital, Nantes
  - Rennes University hospital, Rennes

REFERENCES:
- [Derived] Dumoulin N, Cormier G, Varin S, Coiffier G, Albert JD, Le Goff B, Darrieutort-Laffite C. Factors Associated With Clinical Improvement and the Disappearance of Calcifications After Ultrasound-Guided Percutaneous Lavage of Rotator Cuff Calcific Tendinopathy: A Post Hoc Analysis of a Randomized Controlled Trial. Am J Sports Med. 2021 Mar;49(4):883-891. doi: 10.1177/0363546521992359. PMID 33719606
- [Derived] Darrieutort-Laffite C, Varin S, Coiffier G, Albert JD, Planche L, Maugars Y, Cormier G, Le Goff B. Are corticosteroid injections needed after needling and lavage of calcific tendinitis? Randomised, double-blind, non-inferiority trial. Ann Rheum Dis. 2019 Jun;78(6):837-843. doi: 10.1136/annrheumdis-2018-214971. Epub 2019 Apr 11. PMID 30975645